CLINICAL TRIAL: NCT00312884
Title: Home-HF: a Randomised Controlled Evaluation of Home Telemonitoring of Patients With Heart Failure Recently Discharged From Hospital.
Brief Title: Home-HF: Evaluation of Patients With Heart Failure Using Home Telemonitoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Honeywell HomMed (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006EP001B; 05/Q0411/112
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2007-11

CONDITIONS: Heart Failure
Keywords: telemonitoring; heart failure; randomised; hospitalisation; HomMed
MeSH Terms: conditions — Heart Failure

ARMS (2):
- Usual Care (Active Comparator): Recieved usual hospital and community care
  Interventions: Device: HomMed Telemonitoring System
- Intervention Arm (Experimental): Recieved telemonitoring
  Interventions: Device: HomMed Telemonitoring System

INTERVENTIONS:
Device: HomMed Telemonitoring System — The HomMed telemonitoring system allows for patients to monitor their weight, blood pressure, oxygen saturation and symptoms of dyspnoea on a daily basis from their home

SUMMARY:
This project, using home monitoring for the signs and symptoms of heart failure, aims to empower patients to be actively involved in their care and provide rapid access to healthcare services and advice when needed. The telemonitoring system is easy to use and ensures the accurate transfer of information from the home to the hospital. The information is then screened and if important changes are seen, the patient will be contacted by a heart failure nurse who will offer advice and may arrange a clinic visit or suggest alterations to the medication. The project uses modern technology to provide disease management, links the patient in their home with the hospital and reinforces education and self-care behaviour. This innovative programme will be tested to see if it reduces the risk of re-admission to hospital, reduces anxiety, improves quality of life following a hospital admission for heart failure and whether this represents good value for money in terms of the health benefits it provides.

Hypothesis:

Patients using home telemonitoring of signs and symptoms of heart failure following discharge from hospital with chronic heart failure have a reduced risk of all-cause re-hospitalisation when compared with usual care.

DETAILED DESCRIPTION:
This project, using home monitoring for the signs and symptoms of heart failure, aims to empower patients to be actively involved in their care and provide rapid access to healthcare services and advice when needed. This innovative programme will be tested to see if it reduces the risk of re-admission to hospital. In addition economic evaluation will assess whether this represents good value for money in terms of the health benefits it provides.

After fulfilling the inclusion criteria and being consented into the study, the patients will be randomised into either the control or intervention group in a 1:1 ratio.

Intervention Group:

Prior to hospital discharge the patient and carer/family will be shown how to use the HomMed Telemonitoring equipment. Within two working days of discharge the equipment will be installed in their home by the study nurse who will remind them of its use. They will be provided with a written management plan and advice regarding self-monitoring.They will be asked to monitor signs and symptoms of their disease daily using the HomMed telemonitoring system connected to their home phone line.

The data will be reviewed every working day by a study nurse and examined for variance from the agreed parameters. If clinically significant changes are noted a standard protocol will be used to guide the management.

Control group:

Within two working days of discharge the study nurse will visit patients in the control group and provide them with a written management plan and advice regarding self-monitoring. They will receive usual care for that centre which will consist of a recommendation to visit their GP on hospital discharge and a subsequent review in the outpatient clinic. Informal support offered through the hospital heart failure nurse will continue and this contact will be recorded.

Within both groups the Hospital Anxiety and Depression (HAD) questionnaire, the Minnesota Living with Heart Failure(MLWHF) tool and the Euroqol (EQ-5D) questionnaire will be completed at randomisation, and again at 3 and 6 months following hospital discharge. They will be asked to return completed questionnaires in a pre-paid envelope.

Data on patients' use of healthcare services will be collected from both groups using a combination of retrospective questionnaires and prospective health diaries, which will be returned at 3 and 6 months after randomisation.

Drug optimisation will be assessed through review of medication prescription, and drug utilisation through patient self-report.These data will also be collected at 3 and 6 months.

Patients within both groups will be involved in the study for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class II - IV (i.e. breathlessness at rest or on mild-moderate exercise) at time of randomisation (hospital discharge)
* Proven diagnosis of heart failure, in line with the guidelines for management of chronic heart failure of the European Society of Cardiology or as determined by the cardiologist or physician caring for the patient
* Admission to hospital following a new diagnosis of heart failure or episode of acute decompensation of chronic heart failure
* Home telephone line
* Deemed fit for discharge home by the clinical team

Exclusion Criteria:

* Dementia/confusion which is likely to interfere with the use of the HomMed telemonitoring equipment.
* < 18 years of age
* Lack of home telephone line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Cowie, MD MSc FRCP, Principal Investigator — Imperial College London & Royal Brompton and Harefield Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - West Middlesex University Hospital, Greater London, Middlesex
  - Ealing Hospital, London
  - Hillingdon Hospital, Uxbridge

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Recieved home telemonitoring daily HomMed Telemonitoring System: The HomeMed telemonitoring system allows for patients to monitor their weight, blood pressure, oxygen saturation and symptoms of dyspnoea on a daily basis from their home
- Usual Care: Received usual hospital care with no Telemonitoring
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care
Started | 91 | 91
Completed | 74 | 79
Not Completed | 17 | 12

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Recieved usual follow-up care
- Intervention Arm: Received daily home monitoring
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention Arm | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10.4) | 70 (12.8) | 71 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 59 | 62 | 121
Region of Enrollment [Number; unit: participants]
  United Kingdom | 91 | 91 | 182

OUTCOME MEASURES:

1. Primary Outcome: Days Alive and Outside of Hospital
Description: Days alive and outside of hospital (i.e. not admitted)
Time Frame: From date of randomisation for 180 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 91 | 91
Days | 180 [165 to 180] | 178 [90 to 180]

2. Primary Outcome: Patients Hospitalised (All Cause)
Time Frame: From randomisation date to 180 days
Measure: Number; unit: participants
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 91 | 91
participants | 23 | 33

3. Primary Outcome: Number of Days Spent in Hospital
Time Frame: From randomisation date for 180 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 91 | 91
days | 17 [6 to 25] | 13 [8 to 34]

4. Primary Outcome: Number of Hospitalisations (All Cause)
Time Frame: from randomisation for 180 days
Measure: Number; unit: Number of hospitalisations
Arm/Group | Usual Care | Intervention Arm
Number analyzed (Participants) | 91 | 91
Number of hospitalisations | 39 | 44

ADVERSE EVENTS:
Description: Adverse events were collected without regard for teh specific adverse event term.
Groups:
- Usual Care: Recieved usual hospital care
- Intervention Arm: Recieved telemonitoring daily via the HomMed Telemonitoring System: The HomMed telemonitoring system allows for patients to monitor their weight, blood pressure, oxygen saturation and symptoms of dyspnoea on a daily basis from their home
Arm/Group | Usual Care | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 23/91 | 33/91
Other Adverse Events (participants affected / at risk) | 10/91 | 17/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=91) | Intervention Arm (N=91)
Hospitalisation (Cardiac disorders) | 23 (39) | 33 (44) — All cause hospitalisation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=91) | Intervention Arm (N=91)
Heart Failure Admission (Cardiac disorders) | 10 (16) | 17 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No